CLINICAL TRIAL: NCT06523556
Title: Phase 1b/2 Study of Axatilimab (SNDX-6352) + Azacitidine (AZA) in Advanced Phase MPN, MPN/MDS Overlap or High-Risk CMML
Brief Title: Axatilimab With or Without Azacitidine for the Treatment of Patients With Advanced Phase Myeloproliferative Neoplasms, Myeloproliferative Neoplasm/Myelodysplastic Syndrome Overlap or High Risk Chronic Myelomonocytic Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Uma Borate (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor-Investigator, Uma Borate, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OSU-23442; NCI-2024-05515 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-07-09; First posted 2024-07-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Atypical Chronic Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Myelodysplastic/Myeloproliferative Neoplasm; Recurrent Myelodysplastic/Myeloproliferative Neoplasm; Recurrent Myeloproliferative Neoplasm; Refractory Chronic Myelomonocytic Leukemia; Refractory Myelodysplastic/Myeloproliferative Neoplasm; Refractory Myeloproliferative Neoplasm
MeSH Terms: conditions — Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Chronic; Myelodysplastic-Myeloproliferative Diseases; Myeloproliferative Disorders | interventions — axatilimab; Azacitidine; Specimen Handling; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase I (Axatilimab) (Experimental): Patients receive axatilimab IV over 30 minutes on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. At time of phase Ib completion, patients with clinical improvement may transition to phase II. Patients undergo bone marrow biopsy and aspiration and blood sample collection throughout the study.
  Interventions: Biological: Axatilimab; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy
- Phase II (Axatilimab and azacitidine) (Experimental): Patients receive axatilimab IV over 30 minutes on days 1 and 15 and azacitidine IV over 10-40 minutes or SC on days 1-7 of each cycle. Cycles repeat every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve PR or better may continue for up to 24 total cycles. Patients who achieve less than PR receive 2 additional cycles and, if PR or better is achieved, may complete up to 24 total cycles. Patients undergo bone marrow biopsy and aspiration and blood sample collection throughout the study.
  Interventions: Biological: Axatilimab; Drug: Azacitidine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Other: Survey Administration

INTERVENTIONS:
Biological: Axatilimab — Given IV
  Other Names: Anti-M-CSFR Monoclonal Antibody SNDX-6352; SNDX 6352; SNDX-6352; SNDX6352; UCB6352
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
  Arms: Phase II (Axatilimab and azacitidine)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow biopsy and aspiration
Other: Survey Administration — Ancillary study
  Arms: Phase II (Axatilimab and azacitidine)

SUMMARY:
This phase Ib/II trial tests the best dose of axatilimab and effectiveness of axatilimab with or without azacitidine for the treatment of patients with advanced phase myeloproliferative neoplasms (MPN), myeloproliferative neoplasm/myelodysplastic syndrome (MPN/MDS) overlap or high risk chronic myelomonocytic leukemia (CMML). Axatilimab is an antibody that is cloned from a single white blood cell that is known to be able to recognize cancer cells and block a protein on the surface of the white blood cells that may be involved in cancer cell growth. By blocking the proteins, this may slow or halt the growth of the cancer. Azacitidine is in a class of medications called antimetabolites. It works by stopping or slowing the growth of cancer cells. Giving axatilimab with or without azacitidine may be safe and effective in treating patients with advanced phase MPN, MPN/MDS overlap or high risk CMML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase 2 dose (RP2D) of axatilimab in relapsed or refractory patients with advanced phase MPN, MPN/MDS overlap or high-risk CMML.

II. To evaluate the overall response rate of axatilimab + azacitidine (AZA) in newly diagnosed patients with advanced phase MPN, MPN/MDS overlap or high-risk CMML using Savona response criteria.

SECONDARY OBJECTIVES:

I. Determine the safety and tolerability of axatilimab + azacitidine combination therapy in those with newly diagnosed advanced phase MPN, MPN/MDS overlap or high-risk CMML.

II. Determine the quality of life in patients receiving axatilimab + AZA using a Modified Myeloproliferative Neoplasm Symptom Assessment Form (MPNSAF).

III. Determine the effect of axatilimab + azacitidine on symptom relief which will be measured by transfusion burden (platelet and/or packed red blood cell), time in hospital, and immune related side effects specifically reactivation of tuberculosis (TB), infusion-related reactions, hepatotoxicity, pneumonia, pyrexia, sepsis, shortness of breath (SBO), hemoptysis, periorbital edema, fatigue, and pancreatitis.

EXPLORATORY OBJECTIVES:

I. To assess the pharmacokinetics of axatilimab in combination with AZA. II. To describe the prevalence and trajectories of patients' physical activity during treatment.

III. To perform detailed correlative studies related to genetic, biochemical, and immunologic changes that occur with axatilimab in combination with AZA.

OUTLINE: This is a phase I, dose-escalation study of axatilimab followed by a phase II study.

PHASE I: Patients receive axatilimab intravenously (IV) over 30 minutes on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. At time of phase Ib completion, patients with clinical improvement may transition to phase II. Patients undergo bone marrow biopsy and aspiration and blood sample collection throughout the study.

PHASE II: Patients receive axatilimab IV over 30 minutes on days 1 and 15 and azacitidine IV over 10-40 minutes or subcutaneously (SC) on days 1-7 of each cycle. Cycles repeat every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve partial response (PR) or better may continue for up to 24 total cycles. Patients who achieve less than PR receive 2 additional cycles and, if PR or better is achieved, may complete up to 24 total cycles. Patients undergo bone marrow biopsy and aspiration and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 30 days and then every 6 months for up to 24 months after last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study
* Age ≥ 18 years at the date of signing the informed consent form (ICF)
* Morphologically confirmed diagnosis of the following based on 2016 World Health Organization (WHO) classification (Arber et al 2016): Phase 1b, patients with relapsed or refractory of any of the following; phase 2, patients with newly diagnosed of any of the following:

  * Chronic myelomonocytic leukemia (CMML), classified as intermediate-2, OR high-risk per the CMML Specific Prognostic Scoring System (CPSS) Molecular Model
  * Atypical chronic myelocytic leukemia (aCML)
  * MDS/MPN unclassified (MDS/MPN-U)
  * Myeloproliferative neoplasm accelerated phase (MPN-AP)
  * MPN-AP requires a previous diagnosis of polycythemia vera (PV), essential thrombocythemia (ET), or primary myelofibrosis (PMF) with intermediate-2 or high risk disease according to International Prostate Symptom Score (IPSS) as well as progression on or failure to respond to at least one line of therapy.
  * Myelodysplastic syndrome/myeloproliferative neoplasm with ring sideroblasts and thrombocytosis (MDS/MPN-RS-T) or MDS/MPN with SF3B1 mutation and thrombocytosis (MDS/MPN-SF3B1-T).
  * Not suitable for immediate myeloablative/intensive chemotherapy based on investigator assessment of age, comorbidities, local guidelines, institutional practice (any or all of these)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 × ULN (except in the setting of isolated Gilbert syndrome)
* Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73m^2 (estimation based on Modification of Diet in Renal Disease [MDRD] formula, by local laboratory)
* Patient is able to communicate with the investigator and has the ability to comply with the requirements of the study procedures
* Women of childbearing potential and men, if not surgically sterilized, should use adequate contraception from 14 days prior to study entry and until 90 days after the last follow-up visit. Adequate contraception is defined as using hormonal contraceptives or an intrauterine device combined with at least 1 of the following forms of contraception: a diaphragm or cervical cap, or a condom

Exclusion Criteria:

* Previous treatment for MPN or MDS/MPN overlap with chemotherapy or other antineoplastic agents including lenalidomide and hypomethylating agent (HMAs) such as decitabine or azacitidine or INQOVI (oral decitabine) (patients who had up to 2 cycles of hypomethylating agents [HMAs] can be included). However, previous treatment with hydroxyurea and/or ruxolitinib is permitted
* Diagnosis of acute myeloid leukemia (AML) including acute promyelocytic leukemia and extra-medullary AML based on WHO 2016 classification (Arber et al 2016)
* Patients who are candidates for myeloablative or intensive chemotherapy treatment or who do not provide consent for this treatment
* History of organ transplant or allogenic hematopoietic stem cell transplant
* Participants with prior malignancy, except:

  * Participants with history of adequately treated malignancy for which no anticancer systemic therapy (namely chemotherapy, radiotherapy or surgery) is ongoing or required during the course of the study.
  * Participants who are receiving adjuvant therapy such as hormone therapy are eligible. However, participants who developed therapy related neoplasms are not eligible
* Previous known allergy/sensitivity to components of axatilimab
* History of acute or chronic pancreatitis
* History of myositis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities | Up to 42 days after the first dose of study medication
  Includes hematologic and non-hematologic toxicities
Overall response rate | Up to 5 years
  The number of participants whose best response (according to the 2006 International Working Group response criteria) over the efficacy analysis period is a complete response or partial response will be tallied to estimate the overall response rate and provide a 95% exact confidence interval, according to the Clopper-Pearson method.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days after end of treatment
  Adverse events will be tabulated by toxicity grade and relationship with study medication and assessed by Common Terminology Criteria for Adverse Events version 5.0.
Quality of life measured by Modified Myeloproliferative Neoplasm Symptom Assessment Form (MPNSAF) | Up to 5 years
  Will be assessed in patients receiving axatilimab + azacitidine (AZA) and will be determined using a Modified Myeloproliferative Neoplasm Symptom Assessment Form (MPNSAF) score. The MPNSAF score has a range from 0 to 100 with 100 representing the highest level of symptom severity. Descriptive statistics, means and standard deviations or medians and ranges will be applied to summarize the MPNSAF score.
Number of platelet transfusions | Up to 5 years
  Will be assessed in patients receiving axatilimab + azacitidine and will be determined by descriptive statistics.
Number of packed red blood cell transfusions | Up to 5 years
  Will be assessed in patients receiving axatilimab + azacitidine and will be determined by descriptive statistics.
Time in hospital | Up to 5 years
  Will be assessed in patients receiving axatilimab + azacitidine and will be determined by descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Uma M Borate, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu